CLINICAL TRIAL: NCT03077178
Title: Evaluation of the Impact of Locoregional Treatment of Soft Tissue Sarcoma on the Functional Status of Patients Aged 70 Years and Over
Brief Title: Impact of Locoregional Treatment of Soft Tissue Sarcoma on Status of Patients Aged 70 Years and Over
Acronym: SARCOLD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IB2016-01
Record Dates: First submitted 2017-02-20; First posted 2017-03-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma Adult
Keywords: Soft Tissue Sarcoma; Surgery; Functional Impact; Elderly Patient; Geriatrics
MeSH Terms: conditions — Sarcoma | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective cohort (Experimental): Geriatric assessment
  Interventions: Procedure: Geriatric assessment

INTERVENTIONS:
Procedure: Geriatric assessment — Geriatric assessment, questionnaire assessment

SUMMARY:
In order to describe functional impact of surgery in elderly patients treated for lower-limb soft-tissue sarcoma, the investigators set up this project which aims to identify prognostic factors among geriatric and functional assessment.

DETAILED DESCRIPTION:
This is a prospective cohort including 100 patients > 70 year-old treated by surgery for lower-limb soft-tissue sarcoma. Data on clinical and geriatric characteristics of the patient as well as functional and quality of life assessment will be collected among patient participation (3 years). Primary endpoint is to describe evaluation of the Impact of Locoregional Treatment of Soft Tissue Sarcoma on the Functional Status.

ELIGIBILITY:
Inclusion Criteria:

1. Aged more than 70 years,
2. Soft tissue sarcoma histologically proven,
3. Sarcoma of the soft tissues of the lower limbs,
4. Operable disease (first-line treatment or neo-adjuvant therapy),
5. ECOG, Performance Status ≤ 2,
6. Decision of surgery validated in Multidisciplinary Consultation Meeting,
7. Reports of the non-opposition documented in the patient file before any procedure specific to the study,
8. Affiliation to system of Social Security (accordance with article L1121-11 of the Code of Public Health).

Exclusion Criteria:

1. Metastatic disease from the onset or relapse
2. Participation in another study involving a similar geriatric assessment.
3. Geographic, familial, social, psychological or psychiatric factors that make the patient incapable of undergoing the study's follow-up and procedures.
4. Persons deprived of liberty or placed under judicial protection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Physical functioning assessment | Change from baseline until 36 months after surgery
  Quality of life questionnaire QLQ-C30

SECONDARY OUTCOMES:
Functional status assessment (TESS) | Change from baseline until 36 months after surgery
  Toronto Extremity salvage score (TESS) Scale
Functional status assessment (MST) | Change from baseline until 36 months after surgery
  Muskuloskeletal Tumor Society (MST) scale
Quality of life assessment QLQ-C30 | Change from baseline until 36 months after surgery
  Quality of life questionnaire QLQ-C30
Quality of life assessment QLQ-EDL-14 | Change from baseline until 36 months after surgery
  Quality of life questionnaire QLQ-EDL-14
Geriatric parameters assessment - G8 | baseline
  G8 (onco-geratic screening score)
Surgical complications | Change from Day 0 until 12 months after surgery
  classification Clavien Dindo
OS | Change from Day 0 until 36 months after surgery
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No